CLINICAL TRIAL: NCT04471363
Title: Cancer Survivors and Their Romantic Partners' Preferences for a Couples-based Physical Activity Intervention: A Needs Assessment Study
Brief Title: Cancer Survivors and Their Romantic Partners' Preferences for a Couples-based Physical Activity
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-1649.cc
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Cancer Diagnosis; Couples

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Specific Exercise Education: This subsample of participants will watch an audio-recorded PowerPoint presentation created by the study team on the benefits of exercise for survivors, caregivers and romantic couples.
  Interventions: Behavioral: Cancer-Specific Exercise education
- Control: All participants will be asked to indicate their exercise knowledge, self-efficacy, beliefs and intentions.

INTERVENTIONS:
Behavioral: Cancer-Specific Exercise education — An audio-recorded PowerPoint presentation created by the study team on the benefits of exercise for survivors, caregivers and romantic couples.
  Groups: Cancer Specific Exercise Education

SUMMARY:
The goal of this research is to explore cancer survivors' and their romantic partners' interest in a couples-based physical activity intervention and whether cancer-specific exercise education influences exercise beliefs and intentions.

DETAILED DESCRIPTION:
This study will assess multiple predictors of couples-based physical activity interest among both survivors and partners including gender, age, current exercise, relationship satisfaction and partner support for exercise. Additionally, this study will include an experimental manipulation in which half of the sample will be randomized to receive cancer-specific exercise education.

ELIGIBILITY:
In order to be eligible, individuals must answer "Yes" to all of the following statements:

* I am a cancer survivor OR I am the romantic partner of a cancer survivor
* I am not currently undergoing chemotherapy, radiation or surgery nor do I have plans to undergo chemotherapy, radiation or a cancer-related surgery in the next 6 months
* I am in a committed, romantic relationship
* I have access to a computer or tablet with internet
* I have an email address that I am willing to share with the study team
* I am at least 18 years of age and less than 90 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are interested in hearing from cancer survivors and romantic partners from diverse backgrounds. This study is open to both active and inactive individuals. Cancer survivors can have had any type of cancer, cancer treatment, or recurrence(s). Further, we are not limiting participation based on time since diagnosis. Romantic partners do not need to be married, co-habituating, or in a relationship for a specific time-period in order to be eligible. Additionally, this study will not exclude couples in which both individuals are cancer survivors. Lastly, while we prefer both partners within a couple participate, we will not exclude individual participation.
Sampling Method: Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Questionnaire to determine predictors | 45 minutes
  All participants will be asked to indicate their exercise knowledge, self-efficacy, beliefs and intentions. Participation in this study will last approximately 45 minutes, and all data will be collected using an on-line Redcap survey. Predictors to be examined are gender, age, current exercise, relationship satisfaction and partner support for exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No